CLINICAL TRIAL: NCT03784209
Title: Automatic Real-time Diagnosis of Gastric Mucosal Disease Using Probe-based Confocal Laser Endomicroscopy With Artificial Intelligence
Brief Title: Automatic Real-time Diagnosis of Gastric Mucosal Disease Using pCLE With Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of QiLu Hospital, Shandong University
Other Study IDs: 2018SDU-QILU-12
Record Dates: First submitted 2018-12-16; First posted 2018-12-21 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Gastric Diseases; Artificial Intelligence; Confocal Laser Endomicroscopy
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — When a gastric mucosal lesion is found using white light endoscopy , endoscopist will observe this lesion using pCLE and then take biopsy for histology examination.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lesions observed by pCLE: pCLE is used to distinguish the suspected lesions detected by white light endoscopy.
  Interventions: Diagnostic Test: The diagnosis of Artificial Intelligence and endoscopist

INTERVENTIONS:
Diagnostic Test: The diagnosis of Artificial Intelligence and endoscopist — When suspected lesion is observed using pCLE, endoscopist and AI will make a diagnosis independently. In addition, the endoscopist can not see the diagnosis of AI.

SUMMARY:
Probe-based confocal laser endomicroscopy (pCLE) is an endoscopic technique that enables real-time histological evaluation of gastric mucosal disease during ongoing endoscopy examination. However this requires much experience, which limits the application of pCLE. The investigators designed a computer-aided diagnosis program using deep neural network to make diagnosis automatically in pCLE examination and contrast its performance with endoscopists.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 80;
* agree to give written informed consent.

Exclusion Criteria:

* Patients under conditions unsuitable for performing CLE including coagulopathy , impaired renal or hepatic function, pregnancy or breastfeeding, and known allergy to fluorescein sodium;
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who receive the upper gastrointestinal tract pCLE examination and screened that fulfill the eligibility criteria at Qilu Hospital, Shandong University will be enrolled into the study
Sampling Method: Non-Probability Sample
Enrollment: 951 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
The diagnosis efficiency of Artificial Intelligence | 24 months
  The primary outcome is to test the diagnostic accuracy, sensitivity, specificity, PPV, NPV of the Artificial Intelligence for diagnosing gastric mucosal disease on real-time pCLE examination.

SECONDARY OUTCOMES:
Contrast the diagnosis efficiency of Artificial Intelligence with endoscopists | 24 months
  The secondary outcome is to compare the diagnosis efficiency (including diagnostic accuracy, sensitivity, specificity, PPV, NPV for diagnosing gastric mucosal disease on real-time pCLE examination) between Artificial Intelligence and endoscopists.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Endoscopic unit of Qilu Hospital Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Liu G, Li G, Li Z, Shao X, Ji R, Ma T, Zhang Y, Su J, Qi Q, Guo J, He Y, Yang X, Li Y, Zuo X. Deep learning-aided optical biopsy achieves whole-chain diagnosis of Correa cascade of gastric cancer: a prospective study. BMC Med. 2025 Sep 30;23(1):527. doi: 10.1186/s12916-025-04310-9. PMID 41029674